CLINICAL TRIAL: NCT03991780
Title: A Phase 2, Pilot Study to Assess the Safety and Efficacy of Fostamatinib in the Treatment of Chronic Active Antibody Mediated Rejection in Renal Transplantation
Brief Title: Fostamatinib in the Treatment of Chronic Active Antibody Mediated Rejection
Acronym: FOSTAMR
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18HH4488; 2018-000027-14 (EudraCT Number)
Record Dates: First submitted 2019-05-01; First posted 2019-06-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Renal Transplant Rejection
Keywords: Renal transplant rejection; donor specific antibody; antibody mediated rejection; spleen tyrosine kinase; fostamatinib
MeSH Terms: interventions — fostamatinib

STUDY DESIGN:
Intervention Model Description: Single centre, not randomised, open label
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fostamatinib (Experimental): All patients will be given treatment with Fostamatinib. The initial treatment dose will be 100mg of Fostamatinib (tablet taken orally) twice daily for 8 weeks. If after 8 weeks the participant has not experienced any side effects and are tolerant of this dose, then the dose will increase to 150mg twice daily. This dose will continue for the duration of the study.
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — All patients will be given treatment with Fostamatinib. The initial treatment dose will be 100mg of Fostamatinib twice daily for 8 weeks. If after 8 weeks the participant has not experienced any side effects and are tolerant of this dose, then the dose will increase to 150mg twice daily. This dose will continue for the duration of the study.
  Other Names: Spleen Tyrosine Kinase Inhibitor, TAVALISSE

SUMMARY:
A Phase 2, Pilot Study to Assess the Safety and Efficacy of Fostamatinib in the Treatment of Chronic Active Antibody Mediated Rejection in Renal Transplantation

DETAILED DESCRIPTION:
The commonest cause of renal transplant failure worldwide is rejection, a process whereby the recipient's immune system recognises the transplant kidney as foreign and attacks it. One common form of rejection is due to the recipient developing antibodies against their kidney transplant. Spleen tyrosine kinase is a molecule present in immune cells which is important in the process of antibody mediated damage. Fostamatinib is a drug which inhibits spleen tyrosine kinase.

This clinical trial will recruit 10 patients who have a renal transplant and a diagnosis of antibody mediated rejection. Patients will be given Fostamatinib for 12 months and will undergo a renal biopsy at 6 months and at a 12 months in order to determine whether the histological signs of antibody mediated rejection have either improved or not progressed.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent prior to any study specific screening procedures.
* Male or female, at least 18 years of age
* Females must be either post-menopausal, surgically sterile (hysterectomy, bilateral salpingectomy or bilateral oophorectomy), or, if of child-bearing potential, must not be pregnant or lactating.
* Patients must be established on tacrolimus maintenance immunosuppression
* A pre-study renal biopsy obtained within 3 months prior to Baseline (Visit 1) will be reviewed by a renal pathologist to ensure subjects meet the following Banff histologic entry criteria: If C4d positive: Microcirculation inflammation score (g+ptc) ≥1 If C4d negative: Microcirculation inflammation score (g+ptc) ≥2 Chronic glomerulopathy (cg) score ≥1b or significant Peritubular Capillary Basement Membrane Multilayering (PTCBML) Chronic tubulo-interstitial scarring ≤50% Glomerular global obsolescence ≤50% Sample must contain at least 7 glomeruli and 1 artery
* Otherwise in stable health as determined by the Investigator based on medical history and laboratory tests during the screening period. See Exclusion Criteria for specific exclusions.
* In the Investigator's opinion, understand the duration of the study (up to 52 weeks), including the requirements for renal biopsies, and has the ability to understand the nature of the study and any hazards of participation and to communicate satisfactorily with the Investigator.

Exclusion Criteria:

* Co-existing Banff Category 4 T-cell mediated rejection
* History of or active, clinically significant, respiratory, gastrointestinal (including pancreatitis), hepatic, neurological, psychiatric, musculoskeletal, genitourinary, dermatological, or other disorder that, in the Investigator's opinion, could affect the conduct of the study or the absorption, metabolism or excretion of the study drug.
* Have had any major cardiovascular event within the 180 days prior to randomisation, including but not limited to: myocardial infarction, unstable angina, cerebrovascular accident, pulmonary embolism, or New York Heart Association Class III or IV heart failure.
* An absolute neutrophil count of < 1,500/μL, Hgb < 9 g/L, ALT or AST of > 1.5x ULN, total bilirubin > 2.0 mg/dL at Baseline (Visit 1).
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea) at Baseline (Visit

  1). The subject may be reassessed after full recovery from the acute gastrointestinal illness.
* Co-existing BK nephropathy or pyelonephritis on screening biopsy.
* Active bacterial, viral or parasitic infections, including tuberculosis. Where CMV viral infection is defined as replicating DNA ≥3000 copies/ml and EBV viral infection is defined as replicating DNA ≥10000 copies/ml.
* Evidence of active or previous invasive fungal infection.
* Positive serologic tests suggestive of active hepatitis B or hepatitis C or hepatitis E(subjects may be included if confirmed hepatitis C recombinant immunoblot assay negative or hepatitis C virus RNA negative [qualitative]) or hepatitis E virus RNA negative by PCR), or subjects with suspected human immunodeficiency virus (HIV).
* Have active malignancy.
* Currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days or 5 half-lives (whichever is longer) from Baseline (Visit 1).
* Are unable or unwilling to follow instructions, including participation in all study assessments and visits.
* Have a history of alcohol or substance abuse that, in the judgment of the Investigator, may impair or risk the subject's full participation in the study.
* Have a condition or be in a situation that the Investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
* Have a known allergy and/or sensitivity to the study drug or its excipients.
* Pregnancy or for women that are sexually active, unable to take highly effective contraception (please see inclusion criteria 3 for more information regarding what classifies as a highly effective contraception method)
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Histological changes of antibody mediated rejection assessed by a histopathologist | 6 months
  Pre treatment and Post treatment renal transplant biopsies will be scored by a histopathologist

SECONDARY OUTCOMES:
Concentration of Protein in urine | 6 months and 12 months
  The Level of proteinuria will be assessed by collected a urine samples which will be sent to the clinical laboratory and the protein/creatinine ratio will be calculated. The normal value of the protein/creatinine ratio should be <10, anything higher than this indicated that the kidney is "leaky" and functioning abnormally. Levels of proteinuria will be compared pre and post treatment
eGFR ( Estimated Glomerular Filtration Rate) assessed by a blood test | 6 months and 12 months
  GFR is Glomerular Filtration Rate and it is a key indicator of renal function. The normal eGFR is 60 or more. If your eGFR is less than 60 for three months or more, your kidneys may not be working well. Th eGFR of participants will be compared pre and post treatment.
Donor specific antibody levels | 6 months and 12 months
  The mean fluorescence intensity (MFI) of donor specific antibody present will be compared pre and post treatment. Each participant will have their Donor specific antibodies measured at baseline pre treatment, this specific antibody or antibodies will be re-measured post treatment and the level (MFI) of the antibody/antibodies will be compared to pre treatment levels.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Tam, MBBChir, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No